CLINICAL TRIAL: NCT05832203
Title: Validation and Effect of the Eats-Up 3.0 Mobile Application With Features of a Balanced and Sustainable Nutrition Diet Recommendation, Healthy Lifestyle, Assessment of Diet Quality and Greenhouse Gas Emission in Adults
Brief Title: Evaluation of Planetary Health Diet Recommendation Using Mobile Application in Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Prof Rina Agustina, MD, PhD, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EARTH
Record Dates: First submitted 2023-03-13; First posted 2023-04-27 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Health Behavior; Overweight and Obesity; Eating Behavior; Calorie Overload
Keywords: Sustainable diet; Adult; Overweight; Obese; Mobile application; Planetary Health Diet
MeSH Terms: conditions — Health Behavior; Overweight; Obesity; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 90 overweight/obese adults will be given counseling on planetary health diet, calorie restriction diet, and healthy lifestyle materials through a mobile app within 6 months
  Interventions: Other: Counseling on planetary health diet with calorie restriction
- Control (Placebo Comparator): 90 overweight/obese adults will be given counseling on balanced nutrition diet, calorie restriction diet, and healthy lifestyle materials through a mobile app within 6 months
  Interventions: Other: Counseling on balanced nutrition diet with calorie restriction

INTERVENTIONS:
Other: Counseling on planetary health diet with calorie restriction — Counselling on planetary healthy diet, calorie restriction diet, and healthy lifestyle through mobile application
  Arms: Intervention
Other: Counseling on balanced nutrition diet with calorie restriction — Counselling on balanced nutrition diet, calorie restriction diet, and healthy lifestyle materials through mobile app
  Arms: Control

SUMMARY:
In recent years, the planetary health diet proposed by the EAT-Lancet Commission has underscored the importance of massive changes to healthy eating on a global scale to prevent environmental degradation. Diet management helps individuals control their food consumption, and this can be supported by the availability of technology through mobile applications. The use of mobile applications considers several aspects such as convenience, comfort, and self-management efficiency in maintaining food consumption. By using an application with the latest features related to diet management, which is equipped with dietary education features, gas emissions, and calculating environmental impacts, it allows users to increase self-awareness to reduce gas emissions from food consumption. Therefore, developing recommendations for a balanced nutritional diet, healthy lifestyle, calculating diet quality, and greenhouse gas emission in one application that is presented in one easy step is an important point in providing comprehensive information for a wider range of potential users. The main objective of this study is to assess the differences in changes in body weight, BMI, waist circumference, and systolic and diastolic blood pressure between the group that was given education on a planetary health diet with calorie restriction and a healthy lifestyle and the group that received education on a balanced diet with calorie restriction and a healthy lifestyle in adults using the 3rd generation of EatsUp mobile application. We will conduct a 24-week intervention for overweight and obese adults.

DETAILED DESCRIPTION:
The EAT-Lancet Commission has proposed a planetary health diet that will improve health, by reducing the burden of non-communicable diseases (NCDs) and will reduce Greenhouse Gas Emissions (GHGE) from food production and consumption globally by up to 80%. The global burden of non-communicable diseases is expected to worsen and the effects of food production on greenhouse gas emissions, nitrogen and phosphorus pollution, loss of biodiversity, and water and land use will reduce the stability of the Earth system. The global food system contributes 19-29% to global greenhouse gas emissions (GHGE) and according to Behrens et al. (2017), the average Indonesian diet produces GHGE of 1.6 KgCO2eq per day. Indonesia, with the characteristics of food consumption depending on the staple food (rice), a slight increase in meat consumption, and the occurrence of obesity in the population of the rich and poor population, shows the early stages of a diet transition. The diet transition effect in developed countries has resulted in an increase in the prevalence of obesity in NCDs, while in developing countries it has caused a double burden of malnutrition. A healthy diet has an appropriate caloric intake and consists of a variety of plant foods, low amounts of animal-sourced foods, unsaturated rather than saturated fats, and small amounts of refined grains, highly processed foods, and added sugars. This study is a randomized clinical trial (RCT) study for overweight and obese adults. The research will be conducted in DKI Jakarta and will consist of 4 (four) stages; screening, recruitment (baseline), providing education, and final data collection (end-line). To find out changes in the provision of education, data will be collected at the beginning of the month and the 6th month (end of the study).

ELIGIBILITY:
Inclusion Criteria:

* 19 - 60 years old
* Female/male
* Domiciled in DKI Jakarta
* Body Mass Index of more than 23
* Having android mobile phone and internet connection
* Having time to participate in the research
* Consists of ordinary adults and health professionals aged 19-65 years in DKI Jakarta

Exclusion Criteria:

* Illiterate
* Breastfeeding mother
* Pregnant women
* Undergoing specific diet program
* Undergoing specific medications related to body weight
* Consuming drugs
* Planning to move residence during the 6 months of the study period
* Not willing to sign informed consent

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | 9, 17, and 24 weeks
  change in Body Mass Index (BMI) obtained from anthropometric measurements (weight (kilograms) and height (meters) converted to Body Mass Index (BMI) score)
Waist circumference | 9, 17, and 24 weeks
  Change in waist circumference obtained from anthropometric measurements.
Systolic blood pressure | 9, 17, 24 weeks
  change in systolic and diastolic blood pressure obtained from blood pressure measurements using calibrated Sphygmomanometer.
Diastolic blood preassure | 9, 17, 24 weeks
  Change in diastolic blood pressure obtained from blood pressure measurements using calibrated sphygmomanometer
Diet Quality | 9, 17, and 24 weeks
  change in diet quality score assessed by Healthy Eating Index (HEI) 2015 scoring system using multiple 24-hour food recall data. The HEI-2015 contains 13 components that sum to a total maximum score of 100 points, the total HEI score is the sum of the adequacy components and moderation components. The closer a set of foods aligns with the Dietary Guidelines for Americans, the higher the HEI score.
Green house gas emissions (GHGE) | 9, 17, and 24 weeks
  change in GHGE score using multiple 24-hour recall data converted to GHGE conversion factor in kilogram of carbon dioxide equivalent per kilogram

SECONDARY OUTCOMES:
Physical activity | 9, 17, and 24 weeks
  Change in physical activity score assessed using The International Physical Activity Questionnaire (IPAQ). The scoring system has three criteria: insufficiently active, minimally Active, and HEPA active.
Sleep quality | 9, 17, and 24 weeks
  Change in sleep quality score assessed using The Pittsburgh Sleep Quality Index (PSQI) questionnaire. The sum of the global PSQI scores ranged from 0 to 21. If Global PSQI score was 5 or less (≤5), considered as good sleep quality, if Global PSQI score was more than 5 (>5), considered as poor sleep quality.
Sel-efficacy | 9, 17, and 24 weeks
  Change in self-efficacy score (nutrition and physical exercise) assessed using the Berlin Risk Appraisal and Health Motivation questionnaire. In each question, the item wording is provided for the three measures. Response format is (1) very uncertain, (2) rather uncertain, (3) rather certain, and (4) very certain. Each response represents points that will be summed up at the end of the question. The bigger the final score, the better the subject's self-efficacy regarding nutrition and physical exercise is.

CONTACTS AND LOCATIONS:
Overall Officials: Rina Agustina, PhD, Principal Investigator — Human Nutrition Research Center, IMERI; Dep of Nutrition, Fac.of Medicine UI
Locations (1):
- Department of Nutrition (FKUI-RSCM); and Human Nutrition Research Center, Indonesian Medical Education Research Institute (HNRC-IMERI) Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tukker A, Goldbohm RA, de Koning A, Verheijden M, Kleijn R, Wolf O, et al. Environmental impacts of changes to healthier diets in Europe. Ecological Economics. 2011 Aug 15;70(10):1776-88.
- [Result] Behrens P, Kiefte-de Jong JC, Bosker T, Rodrigues JFD, de Koning A, Tukker A. Evaluating the environmental impacts of dietary recommendations. Proc Natl Acad Sci U S A. 2017 Dec 19;114(51):13412-13417. doi: 10.1073/pnas.1711889114. Epub 2017 Dec 4. PMID 29203655
- [Result] Popkin BM, Adair LS, Ng SW. Global nutrition transition and the pandemic of obesity in developing countries. Nutr Rev. 2012 Jan;70(1):3-21. doi: 10.1111/j.1753-4887.2011.00456.x. PMID 22221213
- [Result] de Pee S, Hardinsyah R, Jalal F, Kim BF, Semba RD, Deptford A, Fanzo JC, Ramsing R, Nachman KE, McKenzie S, Bloem MW. Balancing a sustained pursuit of nutrition, health, affordability and climate goals: exploring the case of Indonesia. Am J Clin Nutr. 2021 Nov 8;114(5):1686-1697. doi: 10.1093/ajcn/nqab258. PMID 34477830
- [Result] Willett W, Rockstrom J, Loken B, Springmann M, Lang T, Vermeulen S, Garnett T, Tilman D, DeClerck F, Wood A, Jonell M, Clark M, Gordon LJ, Fanzo J, Hawkes C, Zurayk R, Rivera JA, De Vries W, Majele Sibanda L, Afshin A, Chaudhary A, Herrero M, Agustina R, Branca F, Lartey A, Fan S, Crona B, Fox E, Bignet V, Troell M, Lindahl T, Singh S, Cornell SE, Srinath Reddy K, Narain S, Nishtar S, Murray CJL. Food in the Anthropocene: the EAT-Lancet Commission on healthy diets from sustainable food systems. Lancet. 2019 Feb 2;393(10170):447-492. doi: 10.1016/S0140-6736(18)31788-4. Epub 2019 Jan 16. No abstract available. PMID 30660336
- [Result] Abdurahman AA, Bule M, Azadbakhat L, Fallahyekta M, Parouhan A, Qorbani M, Dorosty AR. The association between diet quality and obesity-related metabolic risks. Hum Antibodies. 2020;28(1):1-9. doi: 10.3233/HAB-190387. PMID 31282409
- [Result] Masset G, Soler LG, Vieux F, Darmon N. Identifying sustainable foods: the relationship between environmental impact, nutritional quality, and prices of foods representative of the French diet. J Acad Nutr Diet. 2014 Jun;114(6):862-869. doi: 10.1016/j.jand.2014.02.002. Epub 2014 Apr 4. PMID 24703928
- [Result] Stefani S, Ngatidjan S, Paotiana M, Sitompul KA, Abdullah M, Sulistianingsih DP, Shankar AH, Agustina R. Dietary quality of predominantly traditional diets is associated with blood glucose profiles, but not with total fecal Bifidobacterium in Indonesian women. PLoS One. 2018 Dec 21;13(12):e0208815. doi: 10.1371/journal.pone.0208815. eCollection 2018. PMID 30576336
- [Result] Siregar DAS, Rianda D, Irwinda R, Dwi Utami A, Hanifa H, Shankar AH, Agustina R. Associations between diet quality, blood pressure, and glucose levels among pregnant women in the Asian megacity of Jakarta. PLoS One. 2020 Nov 25;15(11):e0242150. doi: 10.1371/journal.pone.0242150. eCollection 2020. PMID 33237938
- [Result] van de Kamp ME, van Dooren C, Hollander A, Geurts M, Brink EJ, van Rossum C, Biesbroek S, de Valk E, Toxopeus IB, Temme EHM. Healthy diets with reduced environmental impact? - The greenhouse gas emissions of various diets adhering to the Dutch food based dietary guidelines. Food Res Int. 2018 Feb;104:14-24. doi: 10.1016/j.foodres.2017.06.006. Epub 2017 Jun 6. PMID 29433779
- [Result] Ahn JS, Kim DW, Kim J, Park H, Lee JE. Development of a Smartphone Application for Dietary Self-Monitoring. Front Nutr. 2019 Sep 23;6:149. doi: 10.3389/fnut.2019.00149. eCollection 2019. PMID 31608283
- [Result] Choi J, Chung C, Woo H. Diet-Related Mobile Apps to Promote Healthy Eating and Proper Nutrition: A Content Analysis and Quality Assessment. Int J Environ Res Public Health. 2021 Mar 28;18(7):3496. doi: 10.3390/ijerph18073496. PMID 33800531
- [Result] Krebs-Smith SM, Pannucci TE, Subar AF, Kirkpatrick SI, Lerman JL, Tooze JA, Wilson MM, Reedy J. Update of the Healthy Eating Index: HEI-2015. J Acad Nutr Diet. 2018 Sep;118(9):1591-1602. doi: 10.1016/j.jand.2018.05.021. PMID 30146071
- [Result] Rahmi RN, Poolsawad N, Sranacharoenpong K. Environmental Impacts Related to Food Consumption of Indonesian Adults. J Nutr Sci Vitaminol (Tokyo). 2020;66(Supplement):S149-S154. doi: 10.3177/jnsv.66.S149. PMID 33612585
- [Result] David SK, Rafiullah MR. Innovative health informatics as an effective modern strategy in diabetes management: a critical review. Int J Clin Pract. 2016 Jun;70(6):434-49. doi: 10.1111/ijcp.12816. PMID 27238962
- [Result] Alkerwi A. Diet quality concept. Nutrition. 2014 Jun;30(6):613-8. doi: 10.1016/j.nut.2013.10.001. Epub 2013 Oct 14. PMID 24800663
- [Result] Bishwajit G. Nutrition transition in South Asia: the emergence of non-communicable chronic diseases. F1000Res. 2015 Jan 12;4:8. doi: 10.12688/f1000research.5732.2. eCollection 2015. PMID 26834976